CLINICAL TRIAL: NCT07307664
Title: Increasing Germline Genetic Testing for Patients With Cancer
Acronym: gLHS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Josh Peterson (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Josh Peterson, Professor of Biomedical Informatics and Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: gLHS
Record Dates: First submitted 2025-12-26; First posted 2025-12-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Pancreatic Cancer; Conditions or Focus of Study; Hereditary Breast Cancer; Hereditary Colorectal Cancer
Keywords: Genomic Risk; Germline Testing; Hereditary Cancer; Learning Health Systems; Genomic Cancer Risk Assessment; Mainstreaming
MeSH Terms: conditions — Pancreatic carcinoma, familial; Breast Cancer, Familial

STUDY DESIGN:
Intervention Model Description: The clinical intervention the investigators will study is mainstreaming of germline testing by oncology care teams for adult patients with colorectal cancer diagnosed under age 50, female breast cancer diagnosed under age 66, and pancreatic cancer diagnosed at any age. These cancer diagnoses and age ranges follow evidence-based guidelines describing indications for germline testing for these patients (e.g., the National Comprehensive Cancer Network, American Society of Clinical Oncology-Society of Surgical Oncology).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncology physicians and advanced practice providers (Experimental): Clinician members of oncology teams who care for adults with breast, pancreatic, or colorectal cancer will be the target population. We will assess changes in germline test orders for and completion by patients before and after deploying implementation strategies designed to promote testing uptake.
  Interventions: Behavioral: Implementation strategies

INTERVENTIONS:
Behavioral: Implementation strategies — We will deploy different strategy bundles across the clinical sites in three approximate 6-month phases.
  Phase I - Facilitation of provider training, educational materials, and information resources; Patient-facing educational material and information resources Phase II - Audit and feedback report on existing patients; Practice champion support; Optimizing EHR strategies Phase III - EHR tools to facilitate prospective identification of patients, testing, and result reporting

SUMMARY:
Germline testing for hereditary cancer syndromes is underutilized across most health care settings. Using a learning health care approach, the Genomics-enabled Learning Health Systems (gLHS) network aims to evaluate the impact of a suite of implementation strategies to increase germline test ordering by oncology care teams (i.e., mainstreaming) for eligible patients with breast, pancreatic or colorectal cancer. Secondarily, the study will investigate completion of testing by eligible patients, as well as impact on overall rates of germline test ordering in patients with cancer. The network will bundle and deploy different implementation strategies across the clinical sites in three 6-month phases. A maintenance phase after the implementation periods will measure genetic testing rates without any additional implementation strategies to determine persistence of effects. The implementation strategies address clinician-level factors, and thus oncologists and their team members (e.g. advanced practice providers, nurse navigators, case managers) will be the focus of evaluating the impact of implementation strategies. Strategies that will be considered include provider education, audit and feedback reports, facilitation, peer support, and electronic health record (EHR) system optimization to support germline testing. Using the RE-AIM QuEST framework, outcomes will be assessed using mixed methods separately for each eligible cancer type. Data collection from the EHR, other relevant data sources, and qualitative provider feedback will be used to assess ordering and completion of tests and the effect of the implementation strategies on germline testing rates in oncology clinics.

DETAILED DESCRIPTION:
This project seeks to close the acknowledged care gap in genetic testing of hereditary cancer predisposition by evaluating implementation strategies expected to increase guideline-concordant germline genetic testing (referred to in protocol as "germline testing" and defined as testing for inherited gene variants related to cancer) by oncology care teams (i.e., 'mainstreaming', or 'task-shifting' from the traditional genetic consultation referral model). Identification of inherited pathogenic variants in individuals with a cancer diagnosis can have implications for treatment, with targeted therapies. Furthermore, identifying individuals with hereditary risk provides an opportunity for surveillance for early detection of other cancers or risk-reducing procedures. Finally, identifying a pathogenic variant allows for cascade testing in family members, extending these benefits to more individuals. Germline testing for hereditary cancer within current clinical practice is underutilized across most health care settings, even though evidence supports effectiveness to inform clinical care. Mainstreaming is service delivery model that has emerged to improve access to germline testing. It shifts the clinical activities of pre- and post- test germline testing to frontline clinician teams. Here, the investigators will be studying the implementation of mainstreaming throughout the germline testing process, from recognizing patients who are eligible for germline testing to disclosing results for those who opt to test.

The study will assess changes in germline test orders for and completion by patients with cancer who receive care across the clinical sites in the gLHS Network before and after deploying implementation strategies designed to promote testing uptake. There will be three implementation phases followed by a maintenance period. The selected implementation strategies are widely used to improve clinical practice and address barriers previously reported in the literature and documented in participating sites. These strategies will aim to increase mainstreaming of germline testing by oncology teams. Most studies evaluating mainstreaming of germline testing for cancer have been performed in relatively small numbers of patients often at single institutions focusing on outcomes of feasibility and patient and provider satisfaction. Implementation outcomes (e.g., reach, adoption, implementation) precede and impact both service and patient outcomes. Thus, understanding implementation outcomes for mainstreaming of germline testing, as well as contextual factors that are associated with successful implementation, is fundamental to achieving high-quality genetic health care.

ELIGIBILITY:
Inclusion Criteria:

* Oncology care team members (including, but not limited to, oncologists, advanced practice providers, nurse navigators, caring for patients with adult patients with breast cancer, pancreatic cancer or colorectal cancer.

Exclusion Criteria:

* Providers not on the oncology care team

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Germline Genetic Testing Ordered for Breast Cancer Patients | 48 months
  Number of eligible breast cancer patients with germline genetic testing ordered by an oncology care team provider, or associated with an oncology visit, within 7 days of an oncology encounter divided by the number of eligible breast cancer patients seen by the oncology team
Germline Genetic Testing Ordered for Pancreatic Cancer Patients | 48 months
  Number of eligible pancreatic cancer patients with germline genetic testing ordered by an oncology care team provider, or associated with an oncology visit, within 7 days of an oncology encounter divided by the number of eligible pancreatic cancer patients seen by the oncology care team.
Germline Genetic Testing Ordered for Colorectal Cancer Patients | 48 months
  Number of eligible colorectal cancer patients with germline genetic testing ordered by an oncology care team provider, or associated with an oncology visit, within 7 days of an oncology encounter divided by the number of eligible colorectal cancer patients seen by the oncology care team.

SECONDARY OUTCOMES:
Germline Genetic Testing Completed by Breast Cancer Patients | 48 months
  Number of eligible breast cancer patients completing germline testing order that was placed by their oncology care team divided by the number of eligible breast cancer patients with an order placed by the oncology care team determined by EHR data extraction.
Germline Genetic Testing Completed by Pancreatic Cancer Patients | 48 months
  Number of eligible pancreatic cancer patients completing germline testing order that was placed by their oncology care team divided by the number of eligible pancreatic cancer patients with an order placed by the oncology care team determined by EHR data extraction.
Germline Genetic Testing Completed by Colorectal Cancer Patients | 48 months
  Number of eligible colorectal cancer patients completing germline testing order that was placed by their oncology care team divided by the number of eligible colorectal cancer patients with an order placed by the oncology care team determined by EHR data extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Josh F Peterson, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (10):
- United States (10):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Orlando VA Medical Center, Orlando, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Durham VA Medical Center, Durham, North Carolina
  - Salisbury VA Health Care System, Salisbury, North Carolina
  - Geisinger, Danville, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah Health, Salt Lake City, Utah